CLINICAL TRIAL: NCT02334059
Title: Effect of Single Dose Ketamine and Magnesium on Postoperative Pain in Patients Undergoing Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Sanjib D Adhikary, Associate professor, Department of Anesthesiology,, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00001623
Record Dates: First submitted 2014-12-23; First posted 2015-01-08 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Obesity
Keywords: opioid sparing; ketamine; obese; magnesium
MeSH Terms: conditions — Obesity | interventions — Ketamine; Magnesium; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketamine (Active Comparator): Ketamine: 0.5 mg/kg IV dose
  Interventions: Drug: Ketamine; Other: Placebo
- Ketamine plus magnesium (Active Comparator): Ketamine plus magnesium group: 0.5 mg/kg IV dose as well as Magnesium 2 grams IV
  Interventions: Drug: Ketamine plus magnesium
- Placebo (Placebo Comparator): Placebo (normal saline)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine infusion plus placebo infusion of normal saline
  Arms: Ketamine
Drug: Ketamine plus magnesium — Ketamine plus magnesium infusion
  Arms: Ketamine plus magnesium
Other: Placebo — 2 placebo infusions
  Other Names: Normal Saline
  Arms: Ketamine; Placebo

SUMMARY:
Opioid sparing analgesia is extremely important in the post-operative obese population. With more and more obese patients entering the operating room a multi-modal approach to analgesia is crucial. Finding effective alternatives to opioid therapy is the rationale of this proposal. Literature involving ketamine and magnesium in bariatric surgical patients is very sparse.

DETAILED DESCRIPTION:
1. Patient will be identified by surgeon and consented by member of the research team
2. Patient will be randomized to one of three groups on the day of surgery
3. Following securement of the endotracheal tube, the study medication will be administered over 10 minutes via an IV infusion pump.
4. The subject will receive ketamine, ketamine plus magnesium or a placebo.
5. Following surgery, the patient will be taken to the post anesthesia care unit (PACU) and set up with standard ASA monitoring as well as end-tidal CO2 via nasal cannula. A hydromorphone patient controlled analgesia (PCA) pump will be set-up by nursing and given to the patient. Standard dosing of 0.2 mg bolus, every 6 minutes with a maximum 2 mg will be the starting dose as is standard for these patients post-operatively.
6. Primary outcome will be the total amount of hydromorphone used in the first 24 hours post-operatively.

   .

ELIGIBILITY:
Inclusion Criteria:

1. Subjects undergoing laparoscopic sleeve gastrectomy
2. Consenting adults age 18-80
3. ASA II to ASA III
4. Ability to understand and use a PCA
5. Required to be hospitalized for at least 24 hours post-op

Exclusion Criteria:

1. Patient refusal
2. Chronic opiate use (daily opiate use for >3 months)
3. Chronic Kidney disease (Creatinine>2)
4. Known allergy or adverse effect of ketamine, magnesium or hydromorphone
5. Patients with documented psychiatry (Maniac or MDP) history
6. Patient unable to give informed consent
7. Patient with limited or no English fluency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjib Adhikary, MB, BS,MD, Principal Investigator — PSHMC College of Medicine
Locations (1):
- Milton S.Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine | Ketamine Plus Magnesium | Placebo
Started | 37 | 34 | 37
Completed | 37 | 34 | 37
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Ketamine Plus Magnesium | Placebo | Total
Number analyzed (Participants) | 37 | 34 | 37 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.68 (10.82) | 44.15 (11.91) | 39.97 (11.60) | 42.56 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 29 | 85
  Male | 10 | 5 | 8 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 37 | 34 | 37 | 108
BMI [Mean (Standard Deviation); unit: kg/m2] | 47.48 (9.85) | 45.57 (6.73) | 47.37 (8.70) | 46.84 (8.53)
Duration of Surgery [Mean (Standard Deviation); unit: minutes] | 55.14 (8.25) | 67.06 (15.12) | 64.78 (13.23) | 62.19 (13.39)
Pre-operative Pain Score [Mean (Standard Deviation); unit: units on a scale] — Pain Scores will be determined pre-operatively using the Visual Analogue Scale (VAS). The VAS is a 10 point scale, where 0 = no pain and 10 = worst pain a subject has ever felt.
  units on a scale | 0.27 (1.04) | 0.35 (0.95) | 0.41 (1.3) | 0.34 (1.1)
Pre-operative sedation score [Median (Standard Deviation); unit: units on a scale] — Sedation scoring will be determined using the Modified Ramsay Sedation Scale. The Modified Ramsay Sedation Scale is a 6 point scale used to determine alertness, where 1 = patient is awake, anxious, agitated, or restless and 6 = patient with no response to any stimuli (light, noise, or pain). A higher number represents an increased sedative state.
  units on a scale | 2 (0.0) | 1.97 (0.17) | 2 (0.16) | 2 (0.14)
Pre-operative PONV score [Mean (Standard Deviation); unit: units on a scale] — The Pre-Operative PONV score will be determined using the PONV Impact Scale. This scale consists of two questions (rated from 0 to 3) for both questions and the sum of the responses are added for a total PONV score.
  Question 1 asks if an individual has vomited or had any dry retching, where 0 = Not at all, 1 = Once, 2= Twice, and 3= Three or more times.
  Question 2 asks if an individual has experienced a feeling of nausea, where 0 = Not at all, 1 = Sometimes, 2 = Often or most of the time, and 3 = All of the time.
  total score (mean and std deviation) is reported and total ranges from 0-3.
  units on a scale | 0.16 (0.50) | 0.03 (0.17) | 0.14 (0.54) | 0.11 (0.44)

OUTCOME MEASURES:

1. Primary Outcome: Total Hydromorphone Use
Description: Total hydromorphone use in 1st 24 hours post-operatively.
Time Frame: During surgery and 24 hours post-op
Measure: Mean (95% Confidence Interval); unit: mcg/Kg
Arm/Group | Ketamine | Ketamine Plus Magnesium | Placebo
Number analyzed (Participants) | 37 | 34 | 37
mcg/Kg
  Intraoperative | 161.5 [119.6 to 203.3] | 159.6 [109.4 to 209.7] | 195.9 [149.6 to 242.3]
  PACU | 41.9 [20.5 to 63.3] | 47.8 [24.6 to 71.0] | 47.3 [24.1 to 70.5]

2. Secondary Outcome: Pain Scores Using Verbal Analogue Scale (VAS)
Description: Pain scores using VAS scale will be recorded pre-operatively, in the PACU, and every 4 hours until 24 hours post-op. The VAS is a 10 point scale, where 0 = no pain and 10 = the worst pain a subject has ever felt. The highest value 10, indicates an extreme self reported level of pain.
Time Frame: Preoperatively and the 1st 24 hours post-op
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ketamine | Ketamine Plus Magnesium | Placebo
Number analyzed (Participants) | 37 | 34 | 37
units on a scale
  Prior to Surgery | 0.41 [-0.03 to 0.84] | 0.35 [0.02 to 0.68] | 0.27 [-0.08 to 0.62]
  PACU | 5.78 [4.86 to 6.71] | 6.03 [4.86 to 6.78] | 5.95 [4.91 to 6.98]
  4h after surgery | 3.89 [3.20 to 4.57] | 4.29 [3.53 to 5.06] | 4.65 [4.01 to 5.29]
  8h after surgery | 3.67 [3.09 to 4.24] | 3.75 [2.9 to 4.60] | 3.64 [3.08 to 4.20]
  12h after surgery | 3.16 [2.59 to 3.73] | 3.91 [3.28 to 4.53] | 2.69 [2.07 to 3.30]
  16h after surgery | 2.97 [2.3 to 3.64] | 3.64 [2.89 to 4.38] | 3.09 [2.51 to 3.66]
  20h after surgery | 3.22 [2.42 to 4.01] | 4.13 [3.45 to 4.8] | 2.94 [2.36 to 3.53]
  24h after surgery | 3.24 [2.59 to 3.88] | 3.48 [2.81 to 4.15] | 3.33 [2.63 to 4.04]

3. Secondary Outcome: Intraoperative Minimum Alveolar Concentration (MAC) of Desflurane
Description: The average MAC concentration of desflurane will be recorded during the intraoperative period. The Minimum Alveolar Concentration (MAC) of an inhaled anesthetic is the alveolar (or end-expiratory) concentration at which 50% of patients will not show a motor response to a standardized surgical incision.
Time Frame: Intraoperative period
Population: Intraoperative period: Intraoperative Minimum Alveolar Concentration (MAC) of desflurane
Measure: Mean (95% Confidence Interval); unit: Minimal Alveolar Concentration (MAC)
Arm/Group | Ketamine | Ketamine Plus Magnesium | Placebo
Number analyzed (Participants) | 37 | 34 | 37
Minimal Alveolar Concentration (MAC) | 4.05 [3.74 to 4.35] | 4.02 [3.73 to 4.32] | 4.34 [3.98 to 4.71]

ADVERSE EVENTS:
Time Frame: Perioperative time period (within 24 hours) up to 24 hours post surgery
Arm/Group | Ketamine | Ketamine Plus Magnesium | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/34 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/34 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/34 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT02334059/Prot_SAP_000.pdf